CLINICAL TRIAL: NCT06667583
Title: 5p15/ 9q22/ 15q22 Hyperdiploidy and Their Significance in Multiple Myeloma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Gamal Abd El-Nasser, dr dalia gamal, Assiut University
Other Study IDs: Hyperdiploidy in MM Patients
Record Dates: First submitted 2024-10-29; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Multiple Myeloma, Neoplasms
Keywords: Hyperdiploidy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bone Marrow Aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study aims to detect 5p15/ 9q22/ 15q22 hyperdiploidy and thier significance in Multiple Myeloma patients

DETAILED DESCRIPTION:
Multiple myeloma is a malignancy of terminally differentiated B cells(immunoglobulin-producing long lived plasma cells ).Its a Bone Marrow based,multifocal plasma cell neoplasm,Multiple myeloma (MM) is the second most common hematologic malignancy.It is mostly observed in older adults with a median age of 66 to 70 years .The exact etiology of multiple myeloma is unknown. However, frequent alterationsand translocations in the promoter genes, especially chromosome 14, are commonly found in multiple myeloma and likely play a role in disease development.In addition, other oncogenes such as NRAS, KRAS, and BRAF may participate in plasma cell proliferation In the majority of patients,malignant proliferation of plasma cells causes the M protein (abnormal IgG, IgM, or IgA or rarely IgE or IgD) in serum and/or urine. Typical symptoms are hypercalcemia, renal failure, anaemia, or destructive bone lesions ("CRAB") The definition of HD in MM has varied across studies; one study defined HD as numerous chromosomal trisomies and low prevalence of IgH translocations and another as a chromosome count of 48-65, with a gain of at least two odd chromosome, Multiple myeloma can be distinguished into two major subgroups based on the genetic abnormalities that all patients harbor; hyperdiploid MM (≥47 and <75 chromosomes; H-MM) and non-hyperdiploid MM (NH-MM).1 NH-MM is further divided into three subgroups: hypodiploid (≤44 chromosomes), pseudodiploid (45-46 chromosomes) and near tetraploid (>75 chromosomes), H-MM has been defined by multiple chromosomal gains, preferentially of the odd chromosomes 3, 5, 7, 9, 11, 15, 19 and 21.Hyperdiploidy is usually associated with a favourable prognosis.

cytogenetic mutations in MM divided into two classes: primary and secondary. primary mutations that occur during the monoclonal gammopathy of undetermined significance (MGUS) stage, a noncancerous condition that affects plasma cells.The primary mutations typically affect the immunoglobulin genes,the most common trusted Source primary mutation is hyperdiploidy,which causes three chromosomes to develop instead of two, it can be observed in around half of the patients and is considered as a favorable prognostic factor, Secondary mutations occur later in the disease or during its progression.Secondary mutations can also be monosomic, where the mutation causes one member of a chromosome pair to be missing

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed Multiple Myeloma Patients -

Exclusion Criteria:

Patient of Multiple Myeloma who received treatment

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed Multiple Myeloma Patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
detection of 5p15/ 9q22/ 15q22 hyperdiploidy and thier significance in Multiple Myeloma patients | up to 2 yeqrs
  detection of 5p15/ 9q22/ 15q22 hyperdiploidy and thier significance in Multiple Myeloma patients

CONTACTS AND LOCATIONS:
Overall Officials: dalia abd el naser, resident dr, Principal Investigator — Assiut University; Eman Zaki, Professor, Study Director — Assiut University; safia hussein, Lecturer, Study Director — Assiut University; mohammed El nagar, Ass profesor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ravi, G. and Gonsalves, W.I. (2021) Current Diagnosis, Risk Stratification and Treatment Paradigms in Newly Diagnosed Multiple Myeloma. Cancer Treatment and Research Communications, 29, Article ID: 100444 — https://doi.org/10.1016/j.ctarc.2021.100444
- See also: Nassar, S., Taher, A., Spear, R., Wang, F., Madewell, J.E. and Mujtaba, B. (2021) Multiple Myeloma: Role of Imaging in Diagnosis, Staging, and Treatment Response Assessment. Seminars in Ultrasound, CT and MRI, 42, 184-193. — https://doi.org/10.1053/j.sult.2020.08.019
- See also: Abdallah, N., et al. (2020). Cytogenetic abnormalities in multiple myeloma: association with disease characteristics and treatment response. — https://www.nature.com/articles/s41408-020-00348-5